CLINICAL TRIAL: NCT01005121
Title: Colchicine for Diabetic Nephropathy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prof.Avi Livneh (Other Government)
Responsible Party: Sponsor-Investigator, Prof.Avi Livneh, Dept Head, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-09-7369-AL-CTIL
Record Dates: First submitted 2009-10-29; First posted 2009-10-30 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Diabetic Nephropathy
MeSH Terms: conditions — Diabetic Nephropathies | interventions — Colchicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- colchicine (Experimental): patients will receive 2 mg of colchicine daily
  Interventions: Drug: colchicine

INTERVENTIONS:
Drug: colchicine — 2mg, per-os, once daily for six months

SUMMARY:
Patients with diabetic nephropathy and proteinuria, despite maximal anti- hypertensive and anti-glucose treatment, will receive colchicine for six months, 2 mg a day, during which their 24 hour urine protein and renal function tests will be monitored. The investigators' hypothesis is that colchicine will diminish proteinuria and might also help slow down the development of end stage renal failure in the long run.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with DM aging 18+, able to sign an informed consent.
2. 24 hour protein collection between 0.5-6 mg during the last 6 months prior enrollment.
3. Hemoglobin A1c in the range of 6-9%, stable for the last year (0.5±)
4. Creatinine lower than 1.5 mg/dL.
5. Blood pressure lower than 150/90 mmHg on stable anti-hypertensive treatment for at least 3 months.
6. Treated with ACE & ARB, unless contraindicated

Exclusion criteria:

1. Malignancy or significant heart, lung or liver disease.
2. Any GI disease, IBD, malnutrition ( BMI under 18 )
3. Psychiatric disease
4. Any muscle disease, history of rhabdomyelysis, myopathy or myositis.
5. Any disease causing renal injury/proteinuria apart from DM
6. Any inflammatory or autoimmune disease
7. Any infection during the last month.
8. Use of potentially nephrotoxic drugs.
9. Woman in child bearing age that do not use at least one contraceptive device.
10. Pregnant or lactating woman.
11. Participation in another study during the last 3 months.
12. Alcohol or drug abusers
13. Anyone whom the investigators conclude are not appropriate
14. Any patient receiving steroids.
15. Any patient with Colchicine allergy, or treated with the drug during the last two weeks.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-12; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
24 hr urine protein collection | every 2 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba medical center, Tel hashomer, Ramat Gan, Israel